CLINICAL TRIAL: NCT00415597
Title: A Long-Term, Open-Label Safety Study of ALO-01 (Morphine Sulfate Plus Naltrexone Hydrochloride Extended-Release) Capsules in Subjects With Chronic Moderate to Severe Nonmalignant Pain
Brief Title: Study of Embeda (Kadian NT, ALO-01) in Subjects With Chronic Moderate to Severe Nonmalignant Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALO-KNT-302
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Results first posted 2009-10-29 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Pain
Keywords: chronic pain; joint pain; back pain; diabetic peripheral neuropathy; post herpetic neuralgia; ALO-01; Embeda; Chronic Non-Malignant Pain
MeSH Terms: conditions — Pain; Chronic Pain; Arthralgia; Back Pain; Neuralgia, Postherpetic | interventions — morphine, naltrexone combination; Morphine; Naltrexone

ARMS (1):
- ALO-01 (Experimental): Doses given once or twice daily
  Interventions: Drug: ALO-01 (Morphine Sulfate Plus Naltrexone Hydrochloride ER)

INTERVENTIONS:
Drug: ALO-01 (Morphine Sulfate Plus Naltrexone Hydrochloride ER) — capsules, available dosage strengths 20, 30, 40, 50, 60, 80, and 100 mg morphine sulfate with 4% by weight naltrexone hydrochloride given once or twice daily
  Other Names: Embeda

SUMMARY:
Open-Label, Safety Study to evaluate the long-term safety of Kadian NT (ALO-01) administered for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject 18-70 years of age
* Subject agrees to refrain from taking any opioid medications other than study medication during study period.
* History of chronic moderate to severe pain caused by a nonmalignant condition for at least 3 months prior to baseline

Exclusion Criteria:

* Subject has a documented history of allergic reaction or clinically significant intolerance to morphine or other opioids, such that treatment with morphine is contraindicated.
* Subject is pregnant or breast-feeding.
* Subject is receiving chemotherapy, or has an active malignancy of any type or has been diagnosed with cancer within the past three years (excluding squamous or basal cell carcinoma of the skin).
* Subject has a documented history of drug abuse/dependence/misuse or narcotic analgesic abuse/dependence/misuse within five years prior to the Baseline Visit.
* Subject has a Body Mass Index (BMI)>45kg/m2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B. Jones, MD, PharmD, Study Director — Alpharma Pharmaceuticals
Locations (58):
- United States (58):
  - Michael Gibson, MD, Birmingham, Alabama
  - Steven Siwek, MD, Phoenix, Arizona
  - Michael Loes, MD, Phoenix, Arizona
  - Allan Soo, MD, Tempe, Arizona
  - Leah Schmidt, DO, Tucson, Arizona
  - Steve Sitar, MD, Anaheim, California
  - Robert Burton, MD, Anaheim, California
  - Arturo Palencia, MD, Bakersfield, California
  - Adam Karnes, MD, Beverly Hills, California
  - Douglas Haselwood, MD, Fair Oaks, California
  - Steven Croft, MD, Delray Beach, Florida
  - Roberto Rodriquez, MD, Hialeah, Florida
  - Orlando Florete, MD, Jacksonville, Florida
  - Michael Link, MD, Kissimmee, Florida
  - Miguel Trevino, MD, Largo, Florida
  - Diego Torres II, MD, Ormond Beach, Florida
  - Martin Hale, MD, Plantation, Florida
  - Margarita Nunez, MD, St. Petersburg, Florida
  - Mary Stedman, MD, Tampa, Florida
  - Raymond Tidman, MD, Blue Ridge, Georgia
  - Arnold Weil, Marietta, Georgia
  - Marvin Tark, Marietta, Georgia
  - Azazuddin Ahmed, MD, Chicago, Illinois
  - Jenecsis Castro-Skoglund, MD, Peoria, Illinois
  - Steven Elliott, MD, Evansville, Indiana
  - John Peppin, DO, West Des Moines, Iowa
  - Randall Brewer, MD, Shreveport, Louisiana
  - David Miller, MD, North Dartmouth, Massachusetts
  - Adnan Dahdul, MD, Springfield, Massachusetts
  - Rebecca Baumbach, MD, Saginaw, Michigan
  - Mel Lucas, MD, Florissant, Missouri
  - Anthony Margherita, MD, St Louis, Missouri
  - Randale Sechrest, MD, Missoula, Montana
  - John Jacobson, MD, Omaha, Nebraska
  - James Meli, DO, Henderson, Nevada
  - Stephen Miller, MD, Las Vegas, Nevada
  - Vrijendra Kumar, MD, Las Vegas, Nevada
  - Christopher Colopinto, MD, Voorhees Township, New Jersey
  - Barbara McGuire, MD, Albuquerque, New Mexico
  - Arthur Elkind, MD, Mount Vernon, New York
  - Patrick Box, MD, Charlotte, North Carolina
  - Richard Rauck, MD, Winston-Salem, North Carolina
  - Thomas Littlejohn III, MD, Winston-Salem, North Carolina
  - Bruce Corser, MD, Cincinnati, Ohio
  - Gregory Gottschlich, MD, Cincinnati, Ohio
  - Robert Kalb, MD, Toledo, Ohio
  - Tanna Shaw, MD, Oklahoma City, Oklahoma
  - Joseph Dunn, MD, Eugene, Oregon
  - Lawrence Levinson, MD, Tipton, Pennsylvania
  - William Travis Ellison, MD, Greer, South Carolina
  - William Smith, MD, Knoxville, Tennessee
  - Lee Carter, MD, Milan, Tennessee
  - Walter Chase, MD, Austin, Texas
  - Andrew Klymiuk, MD, Richardson, Texas
  - Francis Burch, MD, San Antonio, Texas
  - Suzanne Gazda, MD, San Antonio, Texas
  - Webster Lynn, MD, Salt Lake City, Utah
  - Richard Eckert, MD, Roanoke, Virginia

REFERENCES:
- [Derived] Setnik B, Pixton GC, Webster LR. Safety profile of extended-release morphine sulfate with sequestered naltrexone hydrochloride in older patients: pooled analysis of three clinical trials. Curr Med Res Opin. 2016;32(3):563-72. doi: 10.1185/03007995.2015.1131153. Epub 2016 Jan 26. PMID 26695349
- [Derived] Webster LR, Brewer R, Morris D, Cleveland JM, Setnik B. Opioid titration and conversion in patients receiving morphine sulfate and naltrexone hydrochloride extended release capsules. Postgrad Med. 2011 Sep;123(5):155-64. doi: 10.3810/pgm.2011.09.2471. PMID 21904098
- [Derived] Webster LR, Brewer R, Wang C, Sekora D, Johnson FK, Morris D, Stauffer J. Long-term safety and efficacy of morphine sulfate and naltrexone hydrochloride extended release capsules, a novel formulation containing morphine and sequestered naltrexone, in patients with chronic, moderate to severe pain. J Pain Symptom Manage. 2010 Nov;40(5):734-46. doi: 10.1016/j.jpainsymman.2010.05.004. PMID 21075272

RESULTS

PARTICIPANT FLOW:
Period: Enrollment
Arm/Group | ALO-01
Started | 467
Completed | 465
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Period: Treatment
Arm/Group | ALO-01
Started | 465
Completed | 160
Not Completed | 305
Not completed — Adverse Event | 110
Not completed — Lack of Efficacy | 39
Not completed — Protocol Violation | 67
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 51
Not completed — Lost to Follow-up | 28
Not completed — Drug Screen | 2
Not completed — Administrative | 3
Not completed — Sponsor Decision | 1
Not completed — Multiple Reasons | 1

BASELINE CHARACTERISTICS:
Arm/Group | ALO-01
Number analyzed (Participants) | 465
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 417
  >=65 years | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 51.7 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245
  Male | 220
Brief Pain Inventory (BPI) Average Pain [Mean (Standard Deviation); unit: Units on scale] — All patients reporting a BPI average pain score (over last 24 hours: 0=no pain, 10=worst pain) at baseline
  Units on scale | 6.0 (1.67)

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Treatment Emergent Adverse Events
Description: Number of subjects with adverse events (any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the product whether or not related to the product).
Time Frame: up to 12 months
Population: Patients treated with study drug
Measure: Number; unit: participants
Arm/Group | ALO-01
Number analyzed (Participants) | 465
participants | 378

2. Secondary Outcome: Mean Percent Change From Baseline to 12 Weeks in Brief Pain Inventory Score (BPI) of Average Pain
Description: Percent change in pain intensity scale. Average pain intensity over last 24 hours rated at each visit from 0=no pain to 10=worst pain.
Time Frame: 12 weeks
Population: Patients with data at Week 12
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | ALO-01
Number analyzed (Participants) | 254
Percent change | -31.3 (37.44)
Statistical Analysis 1: Comparison: ALO-01; Null hypothesis: Percent change from baseline = 0; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Mean Percent Change From Baseline to 52 Weeks in Brief Pain Inventory Score (BPI) of Average Pain
Description: as for outcome 2
Time Frame: 52 weeks
Population: Patients with data at Week 52
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | ALO-01
Number analyzed (Participants) | 162
Percent change | -41.5 (39.28)
Statistical Analysis 1: Comparison: ALO-01; Null hypothesis: Percent change from baseline = 0; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | ALO-01
Serious Adverse Events (participants affected / at risk) | 33/465
Other Adverse Events (participants affected / at risk) | 265/465
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALO-01 (N=465)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Arthritis bacterial (Infections and infestations) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Overdose (insulin) (Injury, poisoning and procedural complications) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Ketosis (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Invertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (1)
Somatoform disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 1 (1)
Hip surgery (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALO-01 (N=465)
Constipation (Gastrointestinal disorders) | 148
Nausea (Gastrointestinal disorders) | 117
Vomiting (Gastrointestinal disorders) | 54
Diarrhoea (Gastrointestinal disorders) | 35
Fatigue (General disorders) | 29
Headache (Nervous system disorders) | 56
Somnolence (Nervous system disorders) | 36
Insomnia (Psychiatric disorders) | 27
Pruritus (Skin and subcutaneous tissue disorders) | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the Sponsor for review. Sponsor may request a delay in publication to allow the filing of patent applications before publication or release. The sponsor can require deletion of Confidential Information or request correction of inaccuracies.